CLINICAL TRIAL: NCT01389102
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of Estradiol Metered-Dose Transdermal Spray (MDTS) in the Treatment of Vasomotor Symptoms in Postmenopausal Women
Brief Title: Estradiol Transdermal Spray in the Treatment of Vasomotor Symptoms
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lumara Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EST-01; NCT00122200 (obsolete NCT alias)
Record Dates: First submitted 2011-07-05; First posted 2011-07-07 (Estimated); Results first posted 2012-06-11 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Hot Flashes
Keywords: Postmenopause; Hot Flashes; Estradiol; Polyestradiol phosphate; Estradiol valerate; Estradiol 3-benzoate; Estradiol 17 beta-cypionate; Estrogens; Hormones; Hormones, Hormone Substitutes; Hormone Antagonists
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Placebo transdermal three 90 μL sprays (Placebo Comparator): Placebo transdermal spray, three 90 μL spray applied to adjacent non-overlapping areas on 1 inner forearm daily for 12 weeks using a blinded applicator
  Interventions: Drug: Placebo transdermal three 90 μL sprays
- Placebo transdermal two 90 μL sprays (Placebo Comparator): Placebo transdermal spray, two 90 μL spray applied to adjacent non-overlapping areas on 1 inner forearm daily for 12 weeks using a blinded applicator
  Interventions: Drug: Placebo transdermal two 90 μL sprays
- Placebo transdermal one 90 μL spray (Placebo Comparator): Placebo transdermal spray, one 90 μL spray applied to 1 inner forearm daily for 12 weeks using a blinded applicator
  Interventions: Drug: Placebo transdermal one 90 μL spray
- Estradiol transdermal three 90 μL sprays (Active Comparator): Estradiol transdermal spray, three 90 μL spray applied to adjacent non-overlapping areas on 1 inner forearm daily for 12 weeks using a blinded applicator
  Interventions: Drug: Estradiol transdermal three 90 μL sprays
- Estradiol transdermal two 90 μL sprays (Active Comparator): Estradiol transdermal spray, two 90 μL spray applied to adjacent non-overlapping areas on 1 inner forearm daily for 12 weeks using a blinded applicator
  Interventions: Drug: Estradiol transdermal spray, two 90 μL sprays
- Estradiol transdermal one 90 μL spray (Active Comparator): Estradiol transdermal spray, one 90 μL spray applied to 1 inner forearm daily for 12 weeks using a blinded applicator
  Interventions: Drug: Estradiol transdermal one 90 μL spray

INTERVENTIONS:
Drug: Estradiol transdermal one 90 μL spray — Estradiol transdermal spray, one 90 μL spray applied to 1 inner forearm daily for 12 weeks using a blinded applicator
  Arms: Estradiol transdermal one 90 μL spray
Drug: Estradiol transdermal spray, two 90 μL sprays — Estradiol transdermal spray, two 90 μL spray applied to adjacent non-overlapping areas on 1 inner forearm daily for 12 weeks using a blinded applicator
  Arms: Estradiol transdermal two 90 μL sprays
Drug: Estradiol transdermal three 90 μL sprays — Estradiol transdermal spray, three 90 μL spray applied to adjacent non-overlapping areas on 1 inner forearm daily for 12 weeks using a blinded applicator
  Arms: Estradiol transdermal three 90 μL sprays
Drug: Placebo transdermal two 90 μL sprays — Placebo transdermal spray, two 90 μL spray applied to adjacent non-overlapping areas on 1 inner forearm daily for 12 weeks using a blinded applicator
  Arms: Placebo transdermal two 90 μL sprays
Drug: Placebo transdermal three 90 μL sprays — Placebo transdermal spray, three 90 μL spray applied to adjacent non-overlapping areas on 1 inner forearm daily for 12 weeks using a blinded applicator
  Arms: Placebo transdermal three 90 μL sprays
Drug: Placebo transdermal one 90 μL spray — Placebo transdermal spray, one 90 μL spray applied to 1 inner forearm daily for 12 weeks using a blinded applicator
  Arms: Placebo transdermal one 90 μL spray

SUMMARY:
Estradiol treatment is effective at reducing vasomotor symptoms (eg hot flushes) in postmenopausal women. This study will evaluate the safety and efficacy of Evamist.

DETAILED DESCRIPTION:
Multicenter, randomized, double-blind, placebo-controlled trial evaluating different doses of transdermal estradiol delivered by sray to symptomatic postmenopausal women. The endpoints are the reduction in frequency and severity of hot flushes.

ELIGIBILITY:
Inclusion Criteria:

* Post menopausal women,
* Ages 35 or older,
* Frequent moderate to severe hot flushes,
* Qualifying general medical health

Exclusion Criteria:

* Disqualifying gynecological disorders,
* Disqualifying dermatological disorders,
* Disqualifying concurrent conditions

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 454 (Actual)
Dates: Start 2004-12; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (43):
- United States (43):
  - Alabama Clinical Therapeutics, Birmingham, Alabama
  - Costal Clinical Research, Mobile, Alabama
  - Harmony Clinic, Oro Valley, Arizona
  - Hope Research Institute, Phoenix, Arizona
  - Radiant Research, Phoenix, Arizona
  - Radiant Research, Tucson, Arizona
  - NEA Womens Clinic, Jonesboro, Arkansas
  - Arkansas Women's Center, Little Rock, Arkansas
  - Speciality Care for Women, Redding, California
  - Sacramento Research Medical Grp, Sacramento, California
  - Dr. Steven Drosman, San Diego, California
  - Medical Center for Clinical Research, San Diego, California
  - Benchmark Research, San Francisco, California
  - Pacific Clinical Research, Santa Monica, California
  - Diablo Clinical Research, Walnut Creek, California
  - Downtown Women's Health Care, Denver, Colorado
  - South Florida Medical Research, Aventura, Florida
  - Renstar Medical Research, Ocala, Florida
  - Radiant Research, Pinellas Park, Florida
  - Comprehensive Clinical Trials, West Palm Beach, Florida
  - Radiant Research, Atlanta, Georgia
  - Atlanta West Women's Center, Douglasville, Georgia
  - Radiant Research, Chicago, Illinois
  - Benchmark Research, Metairie, Louisiana
  - Clinical Trials Management, Metairie, Louisiana
  - Women's Health Research Ctr., Laurel, Maryland
  - Ridgeview Research, Chaska, Minnesota
  - Meridian Clinical Research, Omaha, Nebraska
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Radiant Research, Cincinnati, Ohio
  - Radiant Research, Columbus, Ohio
  - TriPhase Research, Franklin, Ohio
  - Radiant Research, Mogadore, Ohio
  - PMG-South/OB-Gyn Health Ctr., Medford, Oregon
  - Center for Women's Medicine, Greenville, South Carolina
  - Clinical Research Associates, Nashville, Tennessee
  - Benchmark Research, Austin, Texas
  - Advanced Research Associates, Corpus Christi, Texas
  - Baylor College of Medicine, Houston, Texas
  - Radiant Research, San Antonio, Texas
  - J. Lewis Research, Salt Lake City, Utah
  - University of Eastern Virginia, Norfold, Virginia
  - Tacoma Women's Specialists, Tacoma, Washington

REFERENCES:
- [Derived] Buster JE, Koltun WD, Pascual ML, Day WW, Peterson C. Low-dose estradiol spray to treat vasomotor symptoms: a randomized controlled trial. Obstet Gynecol. 2008 Jun;111(6):1343-51. doi: 10.1097/AOG.0b013e318175d162. PMID 18515518

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 43 physicians' offices, or their affiliated locations, within the United States between 17 December 2004 and 09 March 2006
Pre-assignment Details: Participants underwent a four week screening period to determine eligibility prior to assignment into the study.
Period: Overall Study
Arm/Group | Placebo Transdermal Three 90 μL Sprays | Placebo Transdermal Two 90 μL Sprays | Placebo Transdermal One 90 μL Spray | Estradiol Transdermal Three 90 μL Sprays | Estradiol Transdermal Two 90 μL Sprays | Estradiol Transdermal One 90 μL Spray
Started | 75 | 76 | 77 | 76 | 74 | 76
Completed | 57 | 64 | 58 | 69 | 61 | 68
Not Completed | 18 | 12 | 19 | 7 | 13 | 8
Not completed — Adverse Event | 1 | 3 | 2 | 2 | 2 | 2
Not completed — Hurricane Katrina | 4 | 2 | 3 | 0 | 3 | 1
Not completed — Lost to Follow-up | 4 | 1 | 1 | 2 | 4 | 1
Not completed — Protocol Violation | 0 | 0 | 3 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 7 | 4 | 9 | 2 | 3 | 3
Not completed — Subject Traveling Out of Country | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Subject Moved | 2 | 0 | 1 | 0 | 0 | 0
Not completed — Unavailable due to husband's illness | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Investigator Judgement | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Transdermal Three 90 μL Sprays | Placebo Transdermal Two 90 μL Sprays | Placebo Transdermal One 90 μL Spray | Estradiol Transdermal Three 90 μL Sprays | Estradiol Transdermal Two 90 μL Sprays | Estradiol Transdermal One 90 μL Spray | Total
Number analyzed (Participants) | 75 | 76 | 77 | 76 | 74 | 76 | 454
Age Continuous [Mean (Standard Deviation); unit: years] | 52.0 (6.3) | 52.0 (7.0) | 52.8 (6.9) | 52.3 (5.7) | 52.2 (6.8) | 53.5 (6.8) | 52.7 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 76 | 77 | 76 | 74 | 76 | 454
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in the Number of Moderate to Severe Vasomotor Symptoms Per Day
Description: Patients completed a daily diary to record the number of mild, moderate and number of moderate or severe vasomotor symptoms [hot flushes and sweating] experienced each day.
  Mild, moderate and severe hot flushes and sweating were defined as follows:
  Mild = sensation of heat without sweating Moderate = sensation of heat with sweating, ability to continue activity Severe = sensation of heat with sweating, causing discontinuation of activity
Time Frame: baseline to week 12
Measure: Mean (Standard Deviation); unit: Vasomotor symptoms per day
Arm/Group | Placebo Transdermal Three 90 μL Sprays | Placebo Transdermal Two 90 μL Sprays | Placebo Transdermal One 90 μL Spray | Estradiol Transdermal Three 90 μL Sprays | Estradiol Transdermal Two 90 μL Sprays | Estradiol Transdermal One 90 μL Spray
Number analyzed (Participants) | 75 | 76 | 77 | 76 | 74 | 76
Vasomotor symptoms per day | -5.32 (6.30) | -6.19 (5.77) | -4.76 (5.84) | -8.44 (4.50) | -8.66 (6.65) | -8.10 (4.02)
Statistical Analysis 1: Comparison: Placebo Transdermal Three 90 μL Sprays vs Estradiol Transdermal Three 90 μL Sprays; Test type: Superiority or Other; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: Placebo Transdermal Two 90 μL Sprays vs Estradiol Transdermal Two 90 μL Sprays; Test type: Superiority or Other; p = 0.0099, ANCOVA
Statistical Analysis 3: Comparison: Estradiol Transdermal One 90 μL Spray; Test type: Superiority or Other; p = 0.0004, ANCOVA

2. Primary Outcome: Mean Change the Severity of Moderate to Severe Vasomotor Symptoms
Description: Patients completed a daily diary to record the number of mild, moderate and severe vasomotor symptoms experienced each day.
  Mild, moderate and severe were defined as follows:
  Mild = sensation of heat without sweating Moderate = sensation of heat with sweating, ability to continue activity Severe = sensation of heat with sweating, causing discontinuation of activity Severity of hot flushes was measured on a scale of none = 0, mild = 1, moderate = 2 and severe = 3.
Time Frame: baseline to week 12 (12 weeks)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo Transdermal Three 90 μL Sprays | Placebo Transdermal Two 90 μL Sprays | Placebo Transdermal One 90 μL Spray | Estradiol Transdermal Three 90 μL Sprays | Estradiol Transdermal Two 90 μL Sprays | Estradiol Transdermal One 90 μL Spray
Number analyzed (Participants) | 75 | 76 | 77 | 76 | 74 | 76
Scores on a scale | -0.31 (0.75) | -0.54 (0.89) | -0.26 (0.60) | -1.07 (1.01) | -0.92 (1.01) | -1.04 (1.01)
Statistical Analysis 1: Comparison: Placebo Transdermal Three 90 μL Sprays vs Estradiol Transdermal Three 90 μL Sprays; Test type: Superiority or Other; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: Placebo Transdermal Two 90 μL Sprays vs Estradiol Transdermal Two 90 μL Sprays; Test type: Superiority or Other; p = 0.0406, ANCOVA
Statistical Analysis 3: Comparison: Placebo Transdermal One 90 μL Spray vs Estradiol Transdermal One 90 μL Spray; Test type: Superiority or Other; p < 0.0001, ANCOVA

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Adverse Events will be collected and assessed during each study visit during the 12 week treatment period and any ongoing events will be followed until resolution or stabilization.
Arm/Group | Placebo Transdermal Three 90 μL Sprays | Placebo Transdermal Two 90 μL Sprays | Placebo Transdermal One 90 μL Spray | Estradiol Transdermal Three 90 μL Sprays | Estradiol Transdermal Two 90 μL Sprays | Estradiol Transdermal One 90 μL Spray
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/76 | 1/77 | 3/76 | 1/74 | 3/76
Other Adverse Events (participants affected / at risk) | 13/75 | 18/76 | 12/77 | 21/76 | 29/74 | 21/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Transdermal Three 90 μL Sprays (N=75) | Placebo Transdermal Two 90 μL Sprays (N=76) | Placebo Transdermal One 90 μL Spray (N=77) | Estradiol Transdermal Three 90 μL Sprays (N=76) | Estradiol Transdermal Two 90 μL Sprays (N=74) | Estradiol Transdermal One 90 μL Spray (N=76)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine Prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Impaired Gastric Emptying (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic Obstructive Airways Disease Excerbated (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Transdermal Three 90 μL Sprays (N=75) | Placebo Transdermal Two 90 μL Sprays (N=76) | Placebo Transdermal One 90 μL Spray (N=77) | Estradiol Transdermal Three 90 μL Sprays (N=76) | Estradiol Transdermal Two 90 μL Sprays (N=74) | Estradiol Transdermal One 90 μL Spray (N=76)
Nasopharyngitis (Infections and infestations) | 1 | 2 | 1 | 1 | 3 | 4
Headache (Nervous system disorders) | 7 | 5 | 4 | 8 | 9 | 7
Breast Tenderness (Reproductive system and breast disorders) | 0 | 4 | 0 | 4 | 5 | 4
Nipple Pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 5 | 2
Nausea (Gastrointestinal disorders) | 4 | 1 | 5 | 2 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 2 | 4 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 4 | 1 | 3 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator shall not publish, or seek to publish, either in whole or in part, any results of the Clinical Investigation without the written consent of the Sponsor.